CLINICAL TRIAL: NCT02499523
Title: Prospective Randomised Controlled Monocentric Study on Acetabulum Patient-specific Pin Drilling Guides
Brief Title: Monocentric Study on Acetabulum Patient-specific Pin Drilling Guides
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Materialise (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMAT003
Record Dates: First submitted 2015-07-01; First posted 2015-07-16 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Threonine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- THR with conventional technique (Active Comparator): Use of conventional technique in THR
  Interventions: Procedure: THR with conventional technique
- THR with ACOG (Experimental): THR with Acetabular Cup Orientation Guides (ACOG)
  Interventions: Procedure: THR with Acetabular Cup Orientation Guides (ACOG)

INTERVENTIONS:
Procedure: THR with conventional technique — THR with conventional technique.
  Arms: THR with conventional technique
Procedure: THR with Acetabular Cup Orientation Guides (ACOG) — THR with the ACOG System.
  Other Names: ACOG, Materialise
  Arms: THR with ACOG

SUMMARY:
A prospective, interventional, monocentric, controlled and randomized study will compare a conventional surgical technique to a surgical technique with the assistance of the Acetabular Cup Orientation Guide (ACOG, Materialise) System during total hip replacement (THR).

DETAILED DESCRIPTION:
Background: The Acetabular Cup Orientation Guide(ACOG) System from MATERIALISE NV was developed and is intended to be used as a surgical instrument to assist in the positioning of acetabular cup components intra-operatively using anatomical landmarks of the pelvis that are clearly identifiable on preoperative computed tomography (CT) imaging scans.

Use of ACOG is a relative new technique. ACOG, based on CT imaging data, fit directly into the patient's anatomy and enable primary total hip replacement . Data showing extra benefit of this technique compared to conventional THR technique are not widely available.

Aim: To determine the safety of this new surgical technique compared to conventional THR.

Methods: 30 participants will be randomized to 2 groups. One group will be operated for a THR with the conventional technique and the other group will be operated for a THR with the assistance of the ACOG System. CT imaging will be taken pre and post operatively to measure cup orientation.

ELIGIBILITY:
Inclusion Criteria:

* Is selected to undergo a primary THR
* Informed consent

Exclusion Criteria:

* Is unable to undergo CT imaging of the full pelvis
* Requires surgical treatment within less than 4 weeks of initiation
* Is unable to undergo a THR through a anterolateral approach
* Presents acute/chronic local or systemic infection
* Is allergic to polyamide
* Patient's BMI > 35
* Patients with severe wear of the acetabular rim or other disorders that affect acetabular rim anatomy and bony landmark recognition.Patients exhibiting severe wear.
* Has impaired decision-making capacity
* Is a prisoner
* Is pregnant
* Has metal components that will result in scatter on the CT imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Acetabular cup positioning | 2 Months post-operatively
  Full leg computed tomography pre-operatively and post-operatively. Cup positioning will be recorded in both groups.

SECONDARY OUTCOMES:
Surgery time | 1 day
Acetabular cup size | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Dolhain, Principal Investigator — AZ Monica
Locations (1):
- AZ Monica, Antwerp, Belgium

REFERENCES:
- [Result] Hananouchi T, Saito M, Koyama T, Hagio K, Murase T, Sugano N, Yoshikawa H. Tailor-made surgical guide based on rapid prototyping technique for cup insertion in total hip arthroplasty. Int J Med Robot. 2009 Jun;5(2):164-9. doi: 10.1002/rcs.243. PMID 19248055
- [Result] Hananouchi T, Saito M, Koyama T, Sugano N, Yoshikawa H. Tailor-made Surgical Guide Reduces Incidence of Outliers of Cup Placement. Clin Orthop Relat Res. 2010 Apr;468(4):1088-95. doi: 10.1007/s11999-009-0994-4. Epub 2009 Jul 24. PMID 19629605